CLINICAL TRIAL: NCT02568631
Title: Improving Social Cognition for Adults With Autism Spectrum Disorder by the Serious Game JeStiMulE Versus Classic Video Game Stimulation Not Improving Social Cognition
Brief Title: Improving Social Cognition for Adults With ASD by the Serious Game JeStiMulE Versus Controls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 15-HPNCL-01
Record Dates: First submitted 2015-09-29; First posted 2015-10-06 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Autistic Disorder
Keywords: Autistic Disorder
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- serious game JeStiMulE (Experimental): * Evaluation of the social cognition for adults with autism.
  * The objective of the players of JeStiMulE (Educational Game for Multisensory Stimulation of Children with developmental disorders) will be to end the game after a period of learning and two periods of game (with emotional words and with idiomatic expressions understanding each three modules). The session ends when the module is carried out, what corresponds approximately at 1 am by module, that is 6 sessions of game.
  * Evaluation of the social cognition for adults with autism.
  Interventions: Other: serious game JeStiMulE
- control video game (Placebo Comparator): * Evaluation of the social cognition for adults with autism.
  * The objective of the players of the control video game will be to play 6 sessions of one hour.
  * Evaluation of the social cognition for adults with autism.
  Interventions: Other: control video game

INTERVENTIONS:
Other: serious game JeStiMulE — The objective of JeStiMulE players will be ending the game after a learning period and two playing periods (with emotional words and idioms, which include three modules each). The session ends when the module is completed, which is approximately one hour per module, or 6 sessions of play.
  Arms: serious game JeStiMulE
Other: control video game — The patients will play 6 sessions of one hour with the control video game
  Arms: control video game

SUMMARY:
The serious game "JeStiMulE" (Educational Game for Multisensory Stimulation of Children with developmental disorders), developed by the Autism Resources Center of Nice, was created to teach social cognition including emotion recognition in context, for children and adolescents with autism. In a previous study, JeStiMulE has demonstrated efficacy in a population of young people aged 6-17 years old with high and low levels of autism.

According to the recommendations of the 2011 HAS, disorders of social interactions are the most persistent troubles of the autistic triad in life.

It seems essential to us to be able to offer young adults with autism, rehabilitation methods adapted to their trouble, and to observe whether JeStiMulE could be one of them.

This study researches the effectiveness of the serious game JeStiMulE in the improvement social cognition for adults with autism versus controls.

The main goal is:

- Comparing the improvement in social cognition among adults with autism using the serious game JeStiMulE or not.

Two groups will be formed: a first one of fifteen adults with a diagnosis of autism objectified, this group will use JeStiMulE and will be compared to a control group of adults with autism, using another video game, not aimed to improve social cognition.

The objective of JeStiMulE players will be ending the game after a learning period and two playing periods (with emotional words and idioms, including three modules each). The groups will be matched with their nonverbal IQ through Raven matrices and visual memory tasks (WAIS).

The control group will also be stimulated through a video game, not specialized in improving social cognition.

The primary outcome will be assessed by the emotion recognition at the FEEST of Ekman test: by the number of emotions recognized on faces, compared to the number of emotion presented through this test.

The secondary outcomes will be:

* The rest of social cognition improvement by several tests (the theory of mind with the score of the Tom-15, the intention with the score Sarfati cartoons, empathy with a self-administered questionnaire: EQ / AQ).
* The impact on the quality of life, verbal fluency of emotional words, and the feedback from JeStiMulE players will also be seen as a secondary outcome.

DETAILED DESCRIPTION:
A lot of studies found a deficit in social cognition for individuals with autism, especially in emotions recognition, more precisely the negative emotions. These studies refer to the population of adults with high-functioning autism, but few reports results for low levels.

The serious game "JeStiMulE" (Educational Game for Multisensory Stimulation of Children with developmental disorders), developed by the Autism Resources Center of Nice, was created to teach social cognition including emotion recognition in context, for children and adolescents with autism, by developing a fun game environment; so that children and adolescents with autism spectrum disorder can experience virtual reality in reciprocal social interactions (emotions recognition, emotional gestures, communication, ...). In a previous study, JeStiMulE has demonstrated its efficacy in a population of young people aged 6-17 years old with high and low levels of autism.

According to the recommendations of the 2011 HAS, disorders of social interactions are the most persistent troubles of the autistic triad in life. But, early stimulation offered by educational provision and care has a positive influence on the development of these disorders.

It seems essential to us to be able to offer young adults with autism, rehabilitation methods adapted to their trouble, and to observe whether JeStiMulE could be one of them.

This study researches the effectiveness of the serious game JeStiMulE in the improvement of social cognition for adults with autism versus controls.

The main goal is:

- Comparing the improvement in social cognition among adults with autism using the serious game JeStiMulE or not.

Two groups will be formed: a first group of fifteen adults with a diagnosis of autism objectified. This group will use JeStiMulE and will be compared to a control group of fifteen adults with autism, using another video game, not aimed to improve social cognition.

The objective of JeStiMulE players will be ending the game after a learning period and two playing periods (with emotional words and idioms, which include three modules each). The session ends when the module is completed, which is approximately one hour per module, or 6 sessions of play. The groups will be matched with their nonverbal IQ through Raven matrices and visual memory tasks (WAIS).

The control group will also be stimulated through a video game, not specialized in improving social cognition.

The primary outcome will be assessed by the emotion recognition at the FEEST of Ekman test: by the number of emotions recognized on faces, compared to the number of emotion presented through this test.

The secondary outcomes will be:

- The rest of social cognition improvement by several tests (the theory of mind with the score of the Tom-15, the intention with the score of the Sarfati BD, empathy with a self-administered questionnaire: EQ / AQ).

All these elements will be tested before and after the playing session to assess improvement of social cognition.

- The impact on the quality of life, verbal fluency of emotional words, and the feedback from JeStiMulE players will also be seen as a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Subjects from 18 to 40 years old.
* Diagnosis of autism according to the diagnostic criteria of the DSM 5
* Cognitive level estimated by the matrices of Raven > 6 years amount age
* Compatible verbal level with the realization of the neurocognitive tests estimated by the verbal indication of understanding of the WAIS
* Legal Subjects or guardian having given their informed consent and written;
* Subjects affiliated to the Social Security.

Exclusion Criteria:

* The subjects with unbalanced epilepsy
* The pregnant women

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09-22 (Actual); Primary Completion 2016-09-20 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Change of Emotion recognition | Comparaison at 4 weeks to baseline
  assessed by the emotion recognition at the FEEST of Ekman test: by the number of emotions recognized on faces, compared to the number of emotion presented through this test.

SECONDARY OUTCOMES:
Change of Social cognition | Comparaison at 4 weeks to baseline
  Comparaison at 4 weeks to baseline after playing 6 sessions of one hour of video game Jestimule or control.
  The rest of social cognition improvement by several tests (the theory of the mind with the score of the Tom-15, the intention with the score Sarfati cartoons, empathy with a self-administered questionnaire: EQ / AQ).
Change of impact on quality of life | Comparaison at 4 weeks to baseline
  The impact on quality of life will be evaluated by Vineland test
Impact on the verbal fluency of emotional words (number of words emitted perminute) | Comparaison at 4 weeks to baseline
  The verbal fluence is the number of words emitted per minute at a patient speaking describing a full of imagery scene
Feedback from JeStiMulE players | Comparaison at 4 weeks to baseline
  the feedback from JeStiMulE players will be registered with a questionnary

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie SERRET, MD, Principal Investigator — Fondation Lenval
Locations (3):
- France (3):
  - Fondation Lenval, Nice
  - Hôpital Pasteur - CHU de Nice, Nice
  - Hôpital psychiatrique de Sainte marie, Nice